CLINICAL TRIAL: NCT07186699
Title: Qualitative Study on Detection and Treatment of Non-Small Cell Lung Cancer in Patients With a History of Alcohol or Substance Use Disorder
Brief Title: Qualitative Study on Detection & Tx of NSCLC in Pts w/ a History of Alcohol or SUD
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2N-25-7; NCI-2025-05477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2N-25-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients participate in a semi-structured interview and may participate in a follow-up focus group interview in which preliminary findings are shared and feedback is elicited on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study will attempt to identify social facilitators and barriers to detection and treatment of non-small cell lung cancer in order to learn how a history of substance abuse or alcohol use impacts care for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify social facilitators and barriers to detection and treatment of NSCLC by interviewing a diverse group of patients at Keck, Los Angeles General Medical Center, and Norris Cancer Center with alcohol or substance use disorder history.

OUTLINE: This is an observational study.

Patients participate in a semi-structured interview and may participate in a follow-up focus group interview in which preliminary findings are shared and feedback is elicited on study.

ELIGIBILITY:
Inclusion Criteria:

* * Adults ≥ 18 years of age

  * Histopathologic or cytologic diagnosis of NSCLC
  * Received or receiving curative intent treatment (e.g. surgery, radiation therapy, systemic therapy)
  * History of alcohol use or substance use disorder (other than tobacco use disorder) within the past 10 years, predating the cancer diagnosis
  * Ability to understand and the willingness to sign a written informed consent
  * English or Spanish speaking. Due to need to conduct semi-structured interviews which can develop into free-flowing conversations we need both participant and interviewer to be fluent

Exclusion Criteria:

* Patients with cognitive disability unable to maintain 30-60 minute conversation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC recruited through USC/Norris Comprehensive Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-09-12 (Estimated); Study Completion 2028-09-12 (Estimated)

PRIMARY OUTCOMES:
Thematic saturation | Up to 3 years
  Will use a Danaher framework to approach analyze interview data using NVivo software (NVivo version 11.0, QSR International). Each interview will be analyzed to identify broad themes.

CONTACTS AND LOCATIONS:
Overall Officials: Brooks V Udelsman, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California